CLINICAL TRIAL: NCT03478553
Title: Idiopathic Pulmonary Fibrosis, a Disease Initiated by Mucociliary Dysfunction
Brief Title: The Genetics of Pulmonary Fibrosis
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1147; W81XWH-17-1-0597_1a (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2018-03-12; First posted 2018-03-27 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples including DNA, RNA, Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with IPF
  Interventions: Other: Blood draw; Other: Questionnaire
- Family members without IPF
  Interventions: Other: Blood draw; Other: Questionnaire

INTERVENTIONS:
Other: Blood draw — Blood draw
Other: Questionnaire — Pulmonary Fibrosis Questionnaire

SUMMARY:
This study seeks to screen first degree family members of people with Idiopathic Pulmonary Fibrosis (IPF) for the earliest signs of lung fibrosis.

DETAILED DESCRIPTION:
The purpose of this study is to explore genetic factors associated with the development of pulmonary fibrosis. The investigators aim is to identify and explore genetic loci that affect development of pulmonary fibrosis and also explore related environmental exposures. Idiopathic pulmonary fibrosis (IPF) is one of the interstitial lung diseases under the broader umbrella of idiopathic interstitial pneumonias (IIP). The investigators hypothesize that inherited genetic factors are associated with pulmonary fibrosis. To investigate the genetics of pulmonary fibrosis, the investigators plan to enroll individuals with pulmonary fibrosis and their family members.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old
* Family member diagnosed with IPF

Exclusion Criteria:

- No family member with IPF

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will include up to 20,000 people in the country, both people with IPF and their family members who have never been diagnosed with IPF.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify and explore genetic loci and related environmental exposures in individuals with familial pulmonary fibrosis and their relatives. | Baseline
  The investigators aim is to identify and explore genetic loci that affect development of pulmonary fibrosis and also explore related environmental exposures. Idiopathic pulmonary fibrosis (IPF) is one of the interstitial lung diseases under the broader umbrella of idiopathic interstitial pneumonias (IIP). The investigators hypothesize that inherited genetic factors are associated with pulmonary fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: David A Schwartz, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No